CLINICAL TRIAL: NCT01453504
Title: A Prospective, Randomized, Placebo-controlled, Multicenter, International Phase I/II Trial of RAD001 (Everolimus) in Combination With DHAP as Induction Therapy in Patients With Relapsed or Refractory Hodgkin Lymphoma (HL)
Brief Title: Everolimus in Combination With DHAP in Patients With Relapsed or Refractory Hodgkin Lymphoma
Acronym: HD-R3i
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Peter Borchmann, Prof., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD-R3i
Record Dates: First submitted 2011-10-17; First posted 2011-10-18 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ever-DHAP (Active Comparator): Combination of Everolimus and DHAP
  Interventions: Drug: DHAP; Drug: Everolimus
- Placebo-DHAP (Placebo Comparator)
  Interventions: Drug: DHAP

INTERVENTIONS:
Drug: DHAP — Dexamethasone, Cytarabine, Cisplatin
Drug: Everolimus
  Arms: Ever-DHAP

SUMMARY:
The purpose of this trial is

1. to determine the recommended dose of everolimus for a subsequent Phase II trial
2. to determine the efficacy of everolimus plus DHAP

ELIGIBILITY:
Inclusion Criteria:

* relapsed or refractory Hodgkin Lymphoma
* age 18-60
* histology confirmed relapse

Exclusion Criteria:

* previous therapy with mTOR inhibitor
* current CNS involvement
* other primary malignant disease within the last 3 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2012-08; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity Rate (DLT) | 4 weeks
  Phase I primary outcome measure
Complete Remission Rate (CR) | 4 weeks
  Phase II primary outcome measure

SECONDARY OUTCOMES:
Adverse event rate | 4 weeks
  Phase I secondary outcome measure
Tumor status (assessed by CT) after chemotherapy | 4 weeks
  Phase II secondary outcome measure
Tumor status (assessed by PET) after chemotherapy | 4 weeks
  Phase II secondary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Borchmann, Prof., Study Chair — University of Cologne, German Hodgkin Study Group
Locations (1):
- 1st Dept. of Medicine, Cologne University Hospital, Cologne, Germany

REFERENCES:
- See also: Homepage GHSG — http://www.ghsg.org